CLINICAL TRIAL: NCT04892966
Title: Texture and Color Enhancement Imaging (TXI) Versus Standard White-light (WLI) Colonoscopy for Colorectal Adenoma Detection: a Multicenter, Randomized, Trial
Brief Title: TXI for the Recognition of Adenomas in Colonoscopy
Acronym: TRACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giulio Antonelli, MD, Consultant Gastroenterologist, PhD Student, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TRACK_GA
Record Dates: First submitted 2021-05-03; First posted 2021-05-19 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Polyp

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXI (TXI group) (Experimental): Arm undergoing normal colonoscopy with TXI light
  Interventions: Diagnostic Test: TXI Light Imaging
- WLI (White Light Imaging Group) (Active Comparator): Arm undergoing normal colonoscopy with standard white light
  Interventions: Diagnostic Test: WLI Imaging

INTERVENTIONS:
Diagnostic Test: TXI Light Imaging — Standard Colonoscopy using TXI imaging
  Arms: TXI (TXI group)
Diagnostic Test: WLI Imaging — Standard Colonoscopy using White Light Imaging
  Arms: WLI (White Light Imaging Group)

SUMMARY:
This two parallel arms, randomized, multicenter trial is aimed at evaluating whether TXI is superior to WLI endoscopy in terms of adenoma detection. Secondary aims will be advanced adenoma detection rate, serrated polyp/adenoma detection rate, as well as procedure variables such as withdrawal time.

ELIGIBILITY:
Inclusion criteria:

- All >40 years-old patients undergoing a colonoscopy for primary screening, Faecal Immunochemical Test (FIT) +, post-polypectomy surveillance

Exclusion criteria:

* patients with personal history of colorectal cancer (CRC), or Inflammatory Bowel Disease (IBD).
* Patients affected with Lynch syndrome or Familiar Adenomatous Polyposis.
* patients with inadequate bowel preparation (defined as Boston Bowel Preparation Scale <2 in any colonic segment).
* patients with previous colonic resection.
* patients on antithrombotic therapy, precluding polyp resection.
* patients who were not able or refused to give informed written consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 747 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | 1 year
  the proportion of participants with at least one adenoma (per-patient analysis)

SECONDARY OUTCOMES:
Advanced ADR | 1 year
  as the proportion of participants with at least one advanced adenoma at a per-patient analysis
polyps, adenomas, advanced adenomas and Sessile Serrated Polyps (SSP) per subject | 1 year
  the total number of detected lesions in each group divided by the total number of participants (per polyp analysis)
proximal and flat adenomas detection rate | 1 year
  the total number of detected lesions in each group divided by the total number of participants (per-polyp analysis)
Withdrawal time | 1 year
  Time from the start of the inspection at the cecum and the withdrawal of the colonoscope from the body of the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Dei Castelli, Ariccia, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Antonelli G, Bevivino G, Pecere S, Ebigbo A, Cereatti F, Akizue N, Di Fonzo M, Coppola M, Barbaro F, Walter BM, Sharma P, Caruso A, Okimoto K, Antenucci C, Matsumura T, Zerboni G, Grossi C, Meinikheim M, Papparella LG, Correale L, Costamagna G, Repici A, Spada C, Messmann H, Hassan C, Iacopini F. Texture and color enhancement imaging versus high definition white-light endoscopy for detection of colorectal neoplasia: a randomized trial. Endoscopy. 2023 Dec;55(12):1072-1080. doi: 10.1055/a-2129-7254. Epub 2023 Jul 14. PMID 37451283